CLINICAL TRIAL: NCT02473744
Title: Oedematous Lower Limb Subcutaneous Drainage in Palliative Care
Acronym: DSOPAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I14010 DSOPAL
Record Dates: First submitted 2015-06-08; First posted 2015-06-17 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Edema
Keywords: lower limb edema; subcutaneous drainage; bioelectrical impedance; quality of life
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oedematous lower limb subcutaneous drainage (Experimental): In case of lymphoedema in palliative situation, a subcutaneous drainage can be performed. It is a simple method, easy to use. After topic analgesia, three subcutaneous channels are created and an absorbent pad collects the lymphatic fluid.
  Interventions: Other: subcutaneous drainage

INTERVENTIONS:
Other: subcutaneous drainage — After topic analgesia, three subcutaneous channels are created and an absorbent pad collects the lymphatic fluid.

SUMMARY:
* Background : Edema of lower extremities is a concern ranging from 19 % to 60% of palliative cancer patients. Lymphedema decreases mobility, induces pain, impacts daily activities, esthetic and behavior. Usual treatment is based on diuretics and physiotherapy but is often unsuccessful. In case of conventional treatment failure, in palliative care, subcutaneous drainage can be discussed with the patients. The technique is simple, easy to use but remains off the record. Since 2004, 23 cases were reported with various methods. All the cases reported were undertaken with various technical approaches and efficacy criteria.
* Purpose : Investigator hypothesize that the subcutaneous drainage of edema (SDO) is effective in case of refractory lymphedema of the lower limbs in palliative care and leads to an improvement in QOL in terms of behavioral and autonomy.

DETAILED DESCRIPTION:
• Abstract : In palliative care, lymphedema results from various associations of cancer, hypoalbuminemia, electrolytic disturbances or organ failure. The lymphatic circulation cannot be summarized by the Starling's equation and obstruction cannot explain everything. An interstitial hypothesis underlines the role of the lymphatic pump and edema volume can be a crucial point. The SDO, via the direct liquid removal, can restore the lymphatic pump function. This volumetric effect can explain the long time effect of the SDO and the large range of liquid amount reported in effective SDO. The superficial lymphatic system, in the superficial layer of derma, drains 80 % of lymph flow. In edema, the increased volume leads to the creation of subcutaneous interconnected lacunas. The subcutaneous site for drainage is justified.

After topic anesthesia, three subcutaneous channels are created on the ankle's medial face of the edematous limbs and liquids are absorbed by pads. An additional drainage can be done on the external face of the thigh with liquid collecting bags in bedridden patients.

The study includes clinical examination, total and segmental bioelectrical impedance measured at J0, J4 and on exit or at J7 at the latest and daily weight, umbilic abdominal perimeters and segmental circumferences and QOL evaluation before and after SDO. Bioelectrical impedance is collected from hand-foot, thigh root-foot and under patella calf - foot electrodes. Segmental circumferences are collected at thigh, calf and ankle points identified from bone relief distance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* palliative care patients
* Karnofsky Scale < 50%
* Uni or bilateral lower limb oedema even if associated with lumbar or pelvi-scrotal oedema or ascitis whatever etiology involved (cancer, organ failure, hypoalbuminemia…)
* Effective Social security regimen affiliation
* Signed informed consent

Exclusion Criteria:

* Refusal to take part in the study
* Local anesthesic contraindication
* Infected skin lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Karnofsky's scale | 7 days
  Change in autonomy evaluated by Karnofsky's scale between Day 7 and Day 0

SECONDARY OUTCOMES:
Karnofsky's scale | 4 Days
  Change in autonomy evaluated by Karnofsky's scale between Day 4 and Day 0
The 15th item of the European Organisation for Research and Treatment of Cancer quality of life questionnaires of palliative cancer care patients (EORTC QLQ C15 PAL), | 4 days and 7 days
  Changes in quality of life evaluated by the 15th item of the EORTC QLQ C15 PAL scale between between Day 4/Day 7 and Day 0
Modify Dermatology Life Quality Index (MDLQI) | 4 days and 7 days
  Changes in quality of life related to lymphedema evaluated by the MDLQI between Day 4/Day 7 and Day 0
Verbal numeric scale for pain | 4 days and 7 days
  Changes in pain evaluated by the verbal numeric scale between Day 4/Day 7 and Day 0
Bioelectrical impedance analysis of lower limbs, calves and thighs | 4 days and 7 days
  Changes in bioelectrical impedance of lower limbs, calves and thighs between Day 4/Day 7 and Day 0.
Segmental limb circumferences measurement | 4 days and 7 days
  Variation of the physical measures in time. Changes in segmental limb circumferences between Day 4/Day 7 and Day 0
Abdominal perimeter measurement | 4 days and 7 days
  Variation of the physical measures in time. Changes in abdominal perimeter between Day 4/Day 7 and Day 0
Weight measurement | 4 days and 7 days
  Variation of the physical measures in time. Changes in weight between Day 4/Day 7 and Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand SARDIN, MD, Principal Investigator — University Hospital, Limoges
Locations (7):
- France (7):
  - University hospital, Bordeaux
  - University hospital, Limoges
  - University hospital, Nantes
  - Hospital, Périgueux
  - Joseph Ducuing hospital, Toulouse
  - University hospital, Toulouse
  - Hospital, Valenciennes